CLINICAL TRIAL: NCT04354662
Title: Phase II Study of Toripalimab Combined With Fluorouracil, Leucovorin, Oxaliplatin and Docetaxel (FLOT) in Patients With Locally Advanced, Resectable Gastric Cancer or Gastroesophageal Junction Adenocarcinoma
Brief Title: Toripalimab Combined With FLOT Neoadjuvant Chemotherapy in Patients With Resectable Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gastrim 001
Record Dates: First submitted 2020-04-15; First posted 2020-04-21 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-01

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; Neoadjuvant Chemotherapy; Immunotherapy; Toripalimab; Pathological Remission
MeSH Terms: conditions — Stomach Neoplasms | interventions — toripalimab; Docetaxel; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: This is an open-label, non-randomized, phase II clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab combined with FLOT (Experimental): In the perioperative period, patients with resectable gastric cancer is treated with flot regimen combined with Toripalimab to observe whether the 3-year disease-free survival (DFS) rate, pathological remission rate, R0 resection rate, D2 radical resection rate, 5-year DFS rate and 5-year OS rate could be improved.
  Interventions: Drug: Toripalimab; Drug: Docetaxel; Drug: Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Toripalimab — 240mg d1
  Other Names: JS001
Drug: Docetaxel — 50mg/m2, d1;
Drug: Fluorouracil — 2600 mg/m², d1
Drug: Leucovorin — 200 mg/m², d1
Drug: Oxaliplatin — 85 mg/m², d1

SUMMARY:
Gastric cancer is one of the most common malignant tumors of the digestive tract. Gastric cancer patients diagnosed for the first time in China have a higher proportion of advanced stages and a higher postoperative metastasis rate. Studies have shown that patients with good pathological response after preoperative neoadjuvant therapy (such as tumor regression grade, TRG0 or 1) have a better prognosis. The AIO-FLOT4 study found that preoperative perioperative FLOT chemotherapy not only prolonged the progression-free survival (PFS) time and overall survival (OS) time of patients with advanced gastric cancer, but also increased postoperative pathological remission rate. How to further improve the efficacy of the perioperative treatment plan may be beneficial to improve the long-term survival of gastric cancer patients. Several clinical studies have also confirmed that PD-1 antibody significantly prolongs the life of gastric cancer patients who have failed advanced chemotherapy in the back-line treatment. Thus the investigators plan to conduct this clinical trials to evaluate the safety and efficacy of Toripalimab (PD-1 antibody) combined with FLOT regimen in the perioperative period.The secondary end points included pathological remission rate, resection rate, D2 radical resection rate, 5-year disease-free survival (DFS) rate and 5-year OS rate.

DETAILED DESCRIPTION:
Gastric cancer is one of the most common malignant tumors of the digestive tract, accounting for the second incidence of malignant tumors, and the third mortality factor related to malignant tumors. In China, most patients with gastric cancer diagnosed for the first time are already in the advanced stage, with stage II and III patients accounting for 63%, and the postoperative recurrence rate is higher. Studies have shown that patients with good pathological response after preoperative neoadjuvant therapy (such as TRG0 or 1) have a better prognosis. In recent years, the AIO-FLOT4 study have found that perioperative chemotherapy with FLOT regimen has prolonged the PFS and OS in patients with advanced gastric cancer. It is preferred to recommend perioperative chemotherapy with FLOT regimen for patients with advanced gastric cancer in the NCCN guidelines or Chinese CSCO guidelines. How to further improve the efficacy of the perioperative treatment plan may be beneficial to improve the long-term survival of gastric cancer patients.

Several clinical studies have also confirmed that PD-1 antibody significantly prolongs the life of gastric cancer patients who have failed advanced chemotherapy in the back-line treatment. In the KEYNOTE-059 study, the effectiveness of chemotherapy combined with PD-1 antibody in gastric cancer patients newly treated reached 62%. It is necessary to explore the efficacy of PD-1 antibody combined with FLOT regimen in the perioperative period. Thus the investigators plan to conduct this clinical trials to evaluate the safety and efficacy of Toripalimab (PD-1 antibody) combined with FLOT regimen in the perioperative period.The secondary end points included pathological remission rate, resection rate, D2 radical resection rate, 5-year DFS rate and 5-year OS rate.

ELIGIBILITY:
Inclusion Criteria:

1. locally advanced (>T1) and/or nodal positive (N+) histologically proven adenocarcinoma of the gastric or gastroesophageal junction without distant metastases (M0)
2. no previous surgical resection
3. no previous cytostatic chemotherapy
4. Age > 18 years, no more than 75 years (female and male)
5. Karnofsky Performance Status score of physical condition is 80-100
6. surgical resectability
7. Exclusion of peritoneal carcinomatosis (if clinically suspected) via laparoscopy
8. Leucocytes > 4.000/µl
9. Platelets > 100.000/µl
10. Serum creatinin ≤ 1.5x of normal value, or Creatinin-Clearance > 50 ml/min
11. written informed consent.

Exclusion Criteria:

1. Distant metastasis or local invasion of adjacent organs;
2. Recurrent or residual gastric cancer;
3. Having or having had autoimmune disease;
4. Previous organ transplantation or HIV patients;
5. Allergy or contraindications to Toripalimab, 5- Fluorouracil, Leucovorin, Oxaliplatin, and Docetaxel;
6. Malignant secondary disease;
7. Severe non-surgical disease or acute infection;
8. Peripheral polyneuropathy > NCI grad I;
9. Blood system, liver and kidney function were damaged;
10. Symptomatic brain metastasis;
11. Obvious arrhythmia, myocardial ischemia, severe atrioventricular block, cardiac insufficiency and severe gravity valve disease;
12. Psychotic subjects who are not easy to control;
13. Pregnant or lactating subjects.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-09-26 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
3-year Disease-Free Survival Rate | Up to 3 years
  The primary end point of the study is the effect of perioperative time flot regimen combined with Toripalimab and D2 radical operation on the 3-year disease-free survival time of resectable gastric cancer.
Pathological complete response rate (pCR) | Up to 6 months
  Proportion of patients with gastric cancer who received Toripalimab combined with FLOT regimen after 4 cycles of neoadjuvant therapy and postoperative pathological examination TRG1a

SECONDARY OUTCOMES:
Major pathological (complete and nearly complete) response (MPR) | Up to 6 months
  Proportion of patients with gastric cancer who received Toripalimab combined with FLOT regimen after 4 cycles of neoadjuvant therapy and postoperative pathological examination TRG1a or 1b.
Adverse Events | Up to 6 months
  For any adverse reactions, the researchers refer to the National Cancer Institute (NCI) standard of common toxicity (CTC)
5-year Disease-Free Rate | Up to 5 years
  The proportion of patients with resectable gastric cancer who have no recurrence or metastasis after 5 years of perioperative treatment
5-year Survival Rate | Up to 5 years
  Proportion of patients with resectable gastric cancer who survived 5 years after perioperative treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hongli Li, Dr, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China